CLINICAL TRIAL: NCT07209059
Title: A Single-Center Pilot Study Evaluating the Efficacy and Safety of First-Line Immunochemotherapy With Nivolumab Guided by Interim PET for Stratification and Hazard Minimization in Patients With Advanced Classical Hodgkin Lymphoma (FINISH-HL)
Brief Title: PET-Adapted First-Line Therapy With Nivolumab for Advanced Hodgkin Lymphoma
Acronym: FINISH-HL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2025
Record Dates: First submitted 2025-07-03; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin Lymphoma; Hodgkin Disease; Advanced Hodgkin Lymphoma
Keywords: Classical Hodgkin Lymphoma; Hodgkin Disease; Nivolumab; Immunotherapy; First-line treatment; PET-adapted therapy; Checkpoint inhibitors; ctDNA; Response-adapted treatment; EACOPD; AVD; PD-1 blockade; Circulating tumor DNA
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Single-arm, response-adapted treatment model. All participants receive the same initial induction therapy (Nivolumab + EACOPD-14), followed by PET-guided stratification into de-escalated, continued, or intensified therapy paths. There is no randomization or comparator group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Response-adapted immunochemotherapy (FINISH protocol) (Experimental): All participants receive induction immunochemotherapy with nivolumab and EACOPD-14 (2 cycles). Based on interim PET-CT after 2 cycles:
  1. PET-negative (Deauville 1-3): de-escalated consolidation with Nivolumab + AVD ×2, followed by nivolumab monotherapy ×2
  2. PET-positive (Deauville ≥4): continuation of Nivo-EACOPD-14 ×2 (total 4 cycles).
  2.1. If PET becomes negative after 4 cycles: consolidation with Nivo-EACOPD-14 ×2 2.2. If PET remains positive after 4 cycles: patient is withdrawn from the protocol
  Circulating tumor DNA (ctDNA) is collected at baseline, after 2, 4, and 6 cycles for exploratory molecular response assessment.
  Interventions: Drug: Nivolumab; Other: N-EACOPD-14; Other: N-AVD

INTERVENTIONS:
Drug: Nivolumab — Monoclonal antibody targeting PD-1; administered in combination regimens
  Other Names: Opdivo
Other: N-EACOPD-14 — 14-day regimen. Combination of Nivolumab with Etoposide, Doxorubicin, Cyclophosphamide, Vincristine, Prednisone, and Dacarbazine; given for 2 cycles as initial therapy.
  Other Names: Nivolumab + EACOPD
Other: N-AVD — Combination of Nivolumab with Doxorubicin, Vinblastine, and Dacarbazine; used as de-escalated therapy after negative interim PET (2 cycles).
  Other Names: Nivolumab + AVD

SUMMARY:
This is a single-center, open-label, phase 2 pilot study evaluating the efficacy and safety of a response-adapted first-line treatment strategy for patients with classical Hodgkin lymphoma (cHL) and unfavorable prognostic factors. The FINISH protocol (First-line Immuno-chemotherapy Navigated by Interim PET for Stratification and Hazard minimization In Hodgkin lymphoma) integrates nivolumab into induction therapy and tailors subsequent treatment based on interim PET-CT response. The study also includes exploratory monitoring of circulating tumor DNA (ctDNA) to investigate its role in early response assessment and residual disease detection.

DETAILED DESCRIPTION:
The FINISH study (First-line Immuno-chemotherapy Navigated by Interim PET for Stratification and Hazard minimization In Hodgkin lymphoma) is designed to evaluate a novel personalized treatment strategy for newly diagnosed patients with classical Hodgkin lymphoma (cHL) and advanced-stage or bulky disease. All participants receive initial immunochemotherapy with nivolumab plus EACOPD-14. Treatment is then adapted based on interim PET-CT after two cycles. Patients with a complete metabolic response (Deauville score 1-3) receive de-escalated consolidation with Nivo-AVD followed by nivolumab monotherapy. Patients with inadequate metabolic response undergo continued or intensified therapy based on further PET response.

In addition to clinical and imaging-based endpoints, the study incorporates exploratory monitoring of circulating tumor DNA (ctDNA) at predefined time points. This includes analysis of ctDNA kinetics and correlation with PET response, aiming to develop a molecular framework for response stratification and early detection of residual disease.

The primary goal is to increase treatment efficacy while minimizing long-term toxicity through PET-guided de-escalation and early immunotherapy integration. Safety, feasibility, and molecular response patterns will be analyzed to inform future trials.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to any study-specific procedures
* Histologically confirmed classical Hodgkin lymphoma (cHL)
* Newly diagnosed disease, Ann Arbor stage IIB (bulky), III, or IV
* At least one measurable lesion ≥15 mm in the longest diameter (by CT)
* Age between 18 and 60 years (inclusive)
* ECOG performance status 0-2
* PET-CT performed at baseline
* No prior chemotherapy, radiotherapy, or immunotherapy for lymphoma
* Adequate organ function, including:
* Serum creatinine ≤ 0.2 mmol/L
* Absence of severe cardiac, pulmonary, hepatic, or renal dysfunction
* Ability to comply with the study protocol and scheduled visits

Exclusion Criteria:

* Active hepatitis B or C infection
* Positive test for HIV
* Pregnancy or breastfeeding
* Prior or active autoimmune disease requiring systemic therapy
* Vaccination with a live vaccine within 30 days prior to first nivolumab dose
* History of non-infectious pneumonitis requiring corticosteroids
* Prior malignancy (except for adequately treated basal cell carcinoma or cervical carcinoma in situ)
* Congestive heart failure, unstable angina, recent myocardial infarction, or severe cardiac arrhythmias
* Severe renal impairment (serum creatinine > 0.2 mmol/L), unless lymphoma-related
* Severe hepatic dysfunction, unless directly related to lymphoma
* Severe pneumonia with respiratory failure or hypoxemia not corrected within 2-3 days
* Sepsis or hemodynamic instability
* Life-threatening bleeding events (e.g., gastrointestinal or cerebral hemorrhage)
* Cachexia (total serum protein < 35 g/L), unless due to lymphoma-related liver damage
* Decompensated diabetes mellitus
* Any somatic or psychiatric condition that, in the investigator's judgment, precludes informed consent or study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving complete metabolic response (CMR) after 2 cycles of induction therapy | 4 weeks after treatment initiation
  Complete metabolic response is defined as Deauville score 1-3 on PET-CT after two cycles of Nivolumab + EACOPD-14, assessed per LYRIC criteria.
Time to CMR | Up to 6 cycles (approximately 12-14 weeks)
  Time from first dose of study treatment to the first documentation of complete metabolic response (Deauville 1-3) by PET-CT. If CMR is not achieved, patients are censored at last PET assessment.
Proportion of patients achieving CMR at PET-2, PET-4, and PET-6 | Up to 18 weeks after first dose
  Rate of complete metabolic response (Deauville 1-3) assessed at interim and end-of-treatment PET-CT scans after 2, 4, and 6 cycles of therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  Time from the first dose of study treatment to death from any cause. Patients alive at the time of analysis will be censored at the date of last follow-up.
Progression-Free Survival (PFS) | Up to 24 months
  Time from first dose of treatment to documented disease progression or death, whichever occurs first. Progression is defined according to LYRIC criteria.
Event-Free Survival (EFS) | Up to 24 months
  Time from start of therapy to first documented disease progression, relapse, treatment discontinuation for any reason, or death.
Duration of metabolic response | Up to 24 months
  Time from first PET-defined complete metabolic response (Deauville 1-3) to documented disease progression or relapse.
Overall Response Rate (ORR) at PET-2, PET-4, and PET-6 | PET-2 (Week 4), PET-4 (Week 8), PET-6 (Week 12-14)
  Proportion of patients with complete or partial metabolic response according to LYRIC and Deauville criteria at each time point.
Incidence and severity of treatment-emergent adverse events | From first dose until 90 days after last treatment
  Number and grade of adverse events according to CTCAE v5.0, including immune-related adverse events, reported throughout treatment.

OTHER OUTCOMES:
Change in circulating tumor DNA (ctDNA) concentration during treatment | From Day 0 to end of treatment (approximately 12-14 weeks)
  Quantitative change in ctDNA levels at baseline, after 2 cycles (PET-2), after 4 cycles (PET-4), and at the end of therapy.
Correlation between ctDNA clearance and PET-defined metabolic response | Up to 14 weeks
  Correlation coefficient between ctDNA clearance (yes/no, as determined by NGS assay) and PET response (Deauville 1-3 vs ≥4) at PET-2, PET-4, and PET-6.
Prognostic value of detectable ctDNA at the end of therapy | Up to 24 months
  Kaplan-Meier estimated PFS in patients stratified by ctDNA status (positive vs negative) at end of treatment.
ctDNA-based molecular profile of patients resistant to PD-1 blockade | At baseline and at progression (up to 2 years)
  Detection of specific mutations and clonal dynamics in patients with insufficient response to nivolumab-based therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny E Zvonkov, MD, PhD, Study Director — National Medical Research Center for Hematology
Locations (1):
- National Medical Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No